CLINICAL TRIAL: NCT06482892
Title: A Single Arm Clinical Study Evaluating the Safety, Tolerability, and Efficacy of Multiple Intravenous Administration of TP03HN106 in Patients With Critical Limb Ischemia
Brief Title: TP03HN106 in Patients With Critical Limb Ischemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Talengen Institute of Life Sciences, Shenzhen, P.R. China. (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP03HN106-CLI-IIT
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: TP03HN106

INTERVENTIONS:
Drug: TP03HN106 — During the dose escalation phase, subjects will undergo a dose escalation trial of intravenous injection of TP03HN106 for 5 consecutive days to evaluate the safety and tolerance of the subjects to the injection dose of TP03HN106. The preset initial dose for this experiment is 10U/kg, with gradient doses of 20, 30, 40, and 50U/kg. Observe the subjects receiving the investigational drug for any adverse events (AEs) after daily intravenous injection.
  During the maintenance treatment phase, the subjects will undergo two consecutive treatment courses at the final dose during the dose escalation phase. During each treatment course, subjects will complete the collection of efficacy and safety data for 14 consecutive days of medication (administered every 2 days) and 14 days of discontinuation to evaluate the efficacy and safety of TP03HN106 for subjects with critical limb ischemia.

SUMMARY:
Critical limb ischemia (CLI) is the most severe ischemic stage in peripheral arterial disease (PAD) of the lower limbs, characterized by decreased walking ability, resting pain (lasting for more than 2 weeks), ulcers, and gangrene, which seriously affect the quality of life of patients. Some patients may even face amputation or death. Thrombosis is an important pathological feature of CLI. TP03HN106 can promote thrombolysis, thus having a therapeutic effect on CLI.

ELIGIBILITY:
Inclusion Criteria:

1. When signing the informed consent form, the age should be ≥ 18 years old, regardless of gender;
2. Clinically diagnosed as a patient with Critical limb ischemia, with a Rutherford score of 4-6.
3. Patients who are unable to undergo interventional surgical treatment, or whose previous interventional surgical treatment is ineffective, or who are unwilling to undergo any intervention or surgical treatment, and can only receive conventional antiplatelet and vasodilator drugs (before baseline, antiplatelet and vasodilator drugs must be used for at least 1 week);
4. During the screening period, lower limb artery color ultrasound or lower limb computed tomography angiography (CTA) showed severe stenosis or occlusion of one or more of the common iliac artery, external iliac artery, common femoral artery, superficial femoral artery, popliteal artery, anterior tibial artery, posterior tibial artery, and fibular artery;
5. During the screening period, if there are severe symptoms of lower limb ischemia, meeting any of the following symptoms is sufficient: There is limb rest pain caused by lower limb ischemia, with a disease duration of ≥ 2 weeks, and a VAS score of ≥ 40mm and < 100mm before the first administration; There are limb tissue ulcers caused by lower limb ischemia, with a disease duration of ≥ 2 weeks and limb ulcers (4cm2 ≤ maximum single ulcer area ≤ 25cm2);
6. All subjects with fertility or their spouses must take effective contraceptive measures within 3 months after signing the informed consent form until the completion of the trial;
7. The subjects voluntarily give informed consent and sign an informed consent form (if the subjects and/or their guardians lack reading ability and cannot understand the content of the informed consent, they need to sign together with a fair witness), fully understand the methods and procedures of the experiment, and be able to provide biological samples for testing related indicators in accordance with the experiment requirements.

Exclusion Criteria:

1. Subjects who are known to be allergic to the investigational drug, its excipients, or other human blood products;
2. Patients with limb gangrene greater than 4 cm2;
3. Patients currently suffering from malignant tumor diseases (including those who have previously had malignant tumors but have not been cured);
4. Screening period for patients with liver and kidney failure:
5. Patients who require hemodialysis;
6. Those who have experienced cerebral infarction or cerebral hemorrhage within 3 months prior to signing the informed consent form;
7. During the screening period, subjects with mental illness, obvious mental disorders or epilepsy, including other individuals with no behavioral or cognitive abilities;
8. Hypertensive patients (SBP ≥ 160mmHg and/or DBP ≥ 100mmHg) who cannot be controlled after standardized treatment in the screening period;
9. Individuals who have received fresh plasma, cold precipitates, or blood products containing TP03HN106 components within one month prior to signing the informed consent form;
10. Those who have participated in clinical trials of other drugs or medical devices within one month before signing the informed consent form;
11. Those who have undergone or plan to undergo surgery during the trial period within one month prior to signing the informed consent form;
12. Alcoholism and/or psychoactive substances, drug abusers and dependents (alcoholism standard: the weekly alcohol intake is more than 21 units (male) and 14 units (female) (1 unit=360 mL beer; or 150 mL wine; or 45 mL white spirit);
13. Miscarriage or termination of pregnancy less than 3 months prior to signing the informed consent form, pregnant women and lactating women (currently breastfeeding or not artificially breastfeeding but less than 6 months after delivery);
14. Poor compliance or any other situation that the researcher deems unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall clinical treatment efficacy rate | Day 62
  The VAS score or ulcer area decreases by ≥ 50% compared to baseline when administering day 62, it is considered a clinically effective case.
  The overall clinical efficacy of patient treatment is calculated according to the following formula:
  Overall clinical treatment effectiveness rate=(number of clinically effective cases/total cases) × 100% When the calculated overall clinical success rate is ≥ 70%, the entire clinical trial is considered successful.

SECONDARY OUTCOMES:
Ankle brachial index, ABI | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in ABI of subjects (applicable to patients with ulcers) compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62 ABI:The ratio of ankle artery systolic pressure to ipsilateral brachial artery systolic pressure
TcPO2 | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in TcPO2 of subjects (applicable to patients with ulcers) compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62 TcPO2: transcutaneous oxygen partial pressure
TBI | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in TBI of subjects compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62 TBI: The ratio of toe artery systolic pressure to ipsilateral brachial artery systolic pressure
Overall clinical treatment efficacy rate | Day 6, day 14, day 21, day 34, day 49
  The VAS score or ulcer area decreases by ≥ 50% compared to baseline when administering day 6, day 14, day 21, day 34, day 49, it is considered a clinically effective case.
  The overall clinical efficacy of patient treatment is calculated according to the following formula:
  Overall clinical treatment effectiveness rate=(number of clinically effective cases/total cases) × 100% When the calculated overall clinical success rate is ≥ 70%, the entire clinical trial is considered successful.
Rutherford grading | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in Rutherford grading of subjects compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62

OTHER OUTCOMES:
Coagulation function indicators | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in coagulation function of subjects compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62
Fibrinogen degradation products (FDP) | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in FDP of subjects compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62
Thrombosis 4 items | Baseline, day 6, day 21, day 34, day 49, and day 62
  Changes in thrombosis 4 items of subjects compared to baseline during administration of day 6, day 21, day 34, day 49, and day 62
Computed tomography perfusion (CTP) | Baseline,day 34, day 62
  Changes in blood volume of subjects compared to baseline during administration of day 34 and day 62
Infrared thermal imaging | Baseline,day 34, day 62
  Measure the temperature of the feet and lower leg
Computed tomography perfusion (CTP) | Baseline,day 34, day 62
  Changes in blood flow of subjects compared to baseline during administration of day 34 and day 62

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided